CLINICAL TRIAL: NCT03895346
Title: Mental Training for Adults With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sara W Lazar, Associate Research Scientist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018P002574
Record Dates: First submitted 2019-03-26; First posted 2019-03-29 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Mild Cognitive Impairment; Aging
Keywords: Mindfulness; Meditation; Imaging; MRI
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Mindfulness; Meditation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes assessors will be masked to the group assignment of participants (mindfulness or brain games and puzzles).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Class meeting three times a week for six months, led by a certified mindfulness meditation instructor. Includes instruction and practice on techniques such as breathing, body scan, physical sensations, and yoga.
  Interventions: Behavioral: Mindfulness
- Brain Games and Puzzles (Active Comparator): Class meeting three times a week for six months, led by a qualified instructor. Includes teaching and practice of puzzles such as word searches, crossword puzzles, Sudoku, and KenKen.
  Interventions: Behavioral: Brain Games and Puzzles

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness meditation is a technique of sustained attention and focus, involving preventing the mind from wandering from the meditative object (i.e. breath or body sensations)
  Other Names: Meditation
  Arms: Mindfulness
Behavioral: Brain Games and Puzzles — Intervention will include the instruction and practice of puzzles such as word searches, crossword puzzles, Sudoku, and KenKen.
  Arms: Brain Games and Puzzles

SUMMARY:
This study aims to determine the feasibility and acceptability of conducting a larger randomized clinical trial to test whether individuals with MCI can benefit from mental training programs.

DETAILED DESCRIPTION:
Half of participants will be randomized to a mindfulness group and half to a brain games and puzzles group as forms of mental training. Participants are adults with mild cognitive impairment. Participants will undergo neuropsychological testing, MRI scanning, and qualitative interviews to assess feasibility of conducting a larger randomized clinical trial in a population with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* CDR (clinical dementia rating) of 0.5
* 50-90 years of age
* Able to speak, read, and understand English
* Willing to participate in a 6 month study and undergo 2 MRI scans at Mass General Hospital
* A score suggesting Mild Cognitive Impairment on the Telephone Interview for Cognitive Status (TICS)
* A Mini Mental State Exam adjusted for age and education of 24 to 30
* Stable medications for at least 30 days
* Subjects with well-controlled vascular risk factors such as treated hypertension, treated hyperlipidemia or well-controlled Type II diabetes (glucose levels < 250) will be included.
* Subjects with a history of cerebrovascular problems but have no persistent neurological deficits will be included
* Available for scheduled class times for both study courses
* Able to complete 40 minutes of homework per day during the 6-month course
* CDR (clinical dementia rating) of 0.5

Exclusion Criteria:

* CDR score other than 0.5
* Cardiovascular disease, stroke, congestive heart failure
* Has surgical aneurysm clips, neurostimulator, implanted pumps, metal fragments in eyes, cardiac pacemaker, non-removable nitroglycerin patch, non-MRI compatible cochlear implants, any other non-MRI compatible metal in body
* Has permanent bridgework in upper mouth that could interfere with MRI scan
* Active hematological, renal, pulmonary, endocrine, or hepatic disorders
* Uncontrolled high blood pressure
* Uncontrolled diabetes or insulin-treated diabetes (diabetes that is controlled with no more than one oral medication will be allowed)
* A history of neurological disease or injury, including a history of seizures or significant head trauma (i.e. extended loss of consciousness, bleeding in the brain, Parkinson's disease, stroke)
* Received treatment for cancer within the last year (skin cancer will be allowed as will any cancer more than 2 years since the last treatment)
* Diagnosis of schizophrenia, PTSD, bipolar disorder, or psychotic disorder at any point during lifetime
* Any axis I psychiatric disorder within the last 12 months
* Weighs more than 350 pounds
* Neurological or medical conditions that would interfere with study procedures or confound results, such as conditions that alter cerebral blood flow or metabolism
* Unstable medications or on medications with CNS effects including cholinesterase inhibitors, memantine, and antidepressants
* Use of psychotropic medications within 12 months prior to the study
* Daily use of any medication that alters neural metabolism or blood flow, including chronic use of benzodiazepines, potent CNS penetrant anticholinergic medications (for bladder control or allergies). These medications taken on an as-needed basis (prn) will be allowed. (Over the counter supplements such as Gingko and fish oil will be allowed)
* Any other medications as reviewed by a clinician on a case-by-case basis
* Current regular practice of meditation, yoga, tai chi, Feldenkrais, or other mind-body practice or more than 8 30-minute long mind-body sessions within the last 6 months. Significant prior mind-body experience as determined by the PI based on frequency, duration, recency, and type of practice.
* Claustrophobia
* Any other criteria that will interfere with the subject's participation as determined by study doctor
* Participation in any investigational drug study within 4 weeks of screening.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment feasibility | 6 months
  Number of subjects recruited within 6 months; determine the number of people excluded for each inclusion/exclusion criterion; assessing reasons why eligible people decide not to enroll.
Retention | 6 months
  Remaining in the study for the full duration of all testing time points (yes/no). Quantify the reasons for dropout
Adherence to study protocol | 6 months
  Number of classes attended; number of times the subject practiced prescribed activities at home; number of people who complete each test/assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Lazar, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No